CLINICAL TRIAL: NCT07176156
Title: Evaluation of the Quality of Chat Conversations With the Suicide Helpline Zelfmoordlijn 1813
Acronym: CHATQ-1813
Status: Not yet recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0321
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Suicide Prevention; User Experience; Suicide; Suicidal Ideation
Keywords: suicide prevention; suicide; suicidal ideation; helpline
MeSH Terms: conditions — Suicide Prevention; Suicide; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users of the Zelfmoord1813 chat service: Participants in this study are individuals who contact the chat service of the Zelfmoordlijn 1813 and meet the following criteria:
  * They are 16 years or older
  * They are chatting on their own behalf (not for someone else)
  Participation is entirely voluntary. Before and after the chat conversation, eligible participants are invited to complete a short questionnaire to help researchers understand how the chat affects their emotional state and suicidal thoughts.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational one-time questionnaire study without intervention

SUMMARY:
Suicide remains a serious public health issue in Flanders. Every day, nearly three people die by suicide, and many more attempt it or struggle with suicidal thoughts. The Zelfmoordlijn 1813 is a free and confidential helpline that offers support to people in crisis through phone, chat, and email. In 2024, volunteers had over 23,000 conversations, including nearly 3,000 via chat.

This study, led by the Flemish Centre of Expertise in Suicide Prevention (VLESP) in collaboration with the Centre for Suicide Prevention (CPZ), aims to better understand how people experience the chat service of the Zelfmoordlijn 1813. While previous research has looked at the impact of phone conversations, little is known about how chat conversations affect suicidal thoughts and feelings.

To explore this, people who contact the chat service will be invited to fill out a short questionnaire before and after their conversation. These questionnaires take about 3 minutes each and are completely voluntary. They ask about feelings like hopelessness, crisis, and perceived support, as well as satisfaction with the chat.

The goal is to improve the quality of chat-based crisis support and ensure that people in emotional distress receive the best possible help. This research will help strengthen suicide prevention efforts in Flanders.

ELIGIBILITY:
Inclusion Criteria:

* being at least 16 years of age
* they are chatting on their own behalf (not for someone else)

Exclusion Criteria:

* indication that they do not meet these criteria or are not interested in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants contact the chat service of the helpline Zelfmoordlijn 1813 regarding their suicidality. Participants in the study are recruited via the Zelfmoordlijn 1813's digital chat system. Only chat-users for whom an operator is available at that moment are given the opportunity to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Suicidality | Pre- and post-measurement (immediately before and after the chat conversation)
  Suicidality is assessed using six key indicators: crisis, hopelessness, helplessness, sense of control, intent to die, and perceived social support. These indicators are measured through short online questionnaires administered before and after the chat conversation with the Suicide Line 1813.
  This set of indicators was selected based on prior research into the effectiveness of suicide prevention helplines and core concepts regarding suicidality.

SECONDARY OUTCOMES:
User Satisfaction with the chat conversation. | Post-measurement (immediately after the chat conversation)
  During the post-measurement (immediately after the chat conversation), participants are asked about their satisfaction with the chat, their experiences regarding understanding and any additional comments they wish to share.

OTHER OUTCOMES:
Socio-demographic data | pre-measurement (immediately before the chat conversation)
  Participants will be asked to provide the following demographic information: gender identity and age

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — Flemish Centre of Expertise in Suicide Prevention (Ghent University)
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No